CLINICAL TRIAL: NCT07281170
Title: Xinqiao High-risk Cohort of Diabetes
Brief Title: Xinqiao High-risk Cohort of Diabetes(NICE)
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, China (Other)
Responsible Party: Principal Investigator, Yufan Wang, Director of endocrinology and metabolism department, Shanghai General Hospital, China
Other Study IDs: NICE202508
Record Dates: First submitted 2025-09-17; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Pre Diabetic
Keywords: xinqiao; Pre Diabetic; NICE
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-risk population for diabetes

SUMMARY:
Objective: 1. To systematically screen the high-risk population of diabetes in Xinqiao area, understand the characteristics of early glucose metabolism changes and pancreatic islet function changes in the high-risk population and patients with prediabetes, and establish the first standardized research cohort of high-risk patients and prediabetes patients in Songjiang area.

2. Use CGM monitoring technology to identify the high-risk groups of diabetes and the fluctuation of blood glucose in pre-diabetes, understand their ophthalmology and bone density, observe the annual conversion rate of diabetes, find effective interventions, move forward the management of diabetes, and create a new model for the management of high-risk groups of diabetes.

Research content: Part I: Establishing the first standardized diabetes high-risk population research cohort in Songjiang area The initiative focuses on early screening for high-risk populations with diabetes, shifting the focus downward and advancing prevention measures to detect diabetes at an earlier stage and initiate timely intervention. In Xinqiao District, all high-risk screening cases will undergo medical history documentation, anthropometric measurements, laboratory testing, and regular follow-ups. Standard oral glucose tolerance test (OGTT) methods will be employed to assess fasting blood glucose levels, insulin sensitivity, 2-hour postprandial glucose and insulin levels after a 75g glucose load, and glycated hemoglobin levels. Beyond evaluating glucose metabolism, the screening will also detect other metabolic disorders through routine blood tests including urinalysis, liver/kidney function tests, uric acid levels, lipid profiles, thyroid function, and urine protein/creatinine ratio. The establishment of this premium high-risk screening program in Xinqiao Community will create Songjiang District's first standardized research cohort for diabetes mellitus (DM) and prediabetes patients, carrying significant strategic importance.

Part II: By integrating Clinical Monitoring (CGM) technology with ophthalmological evaluations and bone density ultrasound examinations, we identify characteristics of high-risk diabetic populations and track their disease progression. The CGM system (with auxiliary devices such as the Shansheng Dynamic Glucose Monitoring System) is utilized to monitor blood glucose fluctuations in these individuals. Concurrently, comprehensive ophthalmic assessments-including visual acuity tests, intraocular pressure measurements, fundus photography, OCT scans, OCTA imaging, and SLO examinations-are conducted alongside bone density testing. Annual follow-up evaluations are performed to track clinical outcomes.

Research innovation points and expected results: Research innovation points:

Establish the first standardized research cohort of high-risk and pre-diabetic patients in Songjiang area; move forward the management of diabetes, and create a new management model for high-risk groups of diabetes.

anticipated results

1. Establish a new standardized diabetes high-risk population research cohort with large sample size.
2. Observe the metabolic characteristics, blood glucose fluctuation, ophthalmic conditions and bone density of high-risk groups with diabetes.
3. Find effective interventions to reduce the annual conversion rate of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who provide written informed consen
* Have access to a smartphone
* Hamily history of diabetes or abnormal microglucose level detected once
* Age ≥18 years at the time of consent

Exclusion Criteria:

* Diabetes mellitus
* Any other condition which, in the judgment of the investigator, would make the subject unsuitable for enrollment in the study
* recently surgical histories, trauma, acute cardiovascular complications, or infectious diseases

Ages: 20 Months to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of the high-risk diabetes population who have been living in the Xinqiao community for a long time
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2034-10-20 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of diabetes in high-risk groups during the study | through study completion, an average of 5 year

SECONDARY OUTCOMES:
FPG HbA1c and TIR changes from baseline in high-risk groups | through study completion, an average of 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No